CLINICAL TRIAL: NCT02707315
Title: A Study of Pre-Operative Cyberknife in Patients With Potentially Resectable Pancreas Cancer
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Cooper Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-169
Record Dates: First submitted 2015-10-02; First posted 2016-03-14 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2015-10

CONDITIONS: Pancreas Cancer; Pancreatic Cancer; Adenocarcinoma of the Pancreas; Pancreas Adenocarcinoma; Pancreatic Adenocarcinoma
Keywords: Cyber Knife; CyberKnife; Stereotactic Radiosurgery; CK
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): Chemotherapy:
  Gemcitabine 1000 mg/m2 weekly x 3 on 28 day cycle
  Radiation:
  25 Gy over 5 fractions
  Surgery:
  surgical resection of pancreas
  treatment plan:
  1 cycle of chemotherapy, followed by stereotactic radiosurgery, followed by an additional 6 cycles of chemotherapy or surgical resection
  Interventions: Drug: Gemcitabine; Radiation: Stereotactic Radiosurgery

INTERVENTIONS:
Drug: Gemcitabine
  Other Names: Gemzar
Radiation: Stereotactic Radiosurgery
  Other Names: CyberKnife; Cyber Knife; CK

SUMMARY:
This study is evaluating stereotactic radiosurgery (CyberKnife) plus chemotherapy for the treatment of potentially resectable adenocarcinoma of the pancreas

DETAILED DESCRIPTION:
This study is evaluating the role of neoadjuvant chemotherapy and CyberKnife therapy in increasing the number of patients who are able to successfully undergo definitive surgical management of their pancreatic carcinoma. In addition, we will evaluate the associated therapeutic toxicities and gather data regarding the quality of life indicators at similar time intervals for an improved overall assessment of the effects of this course of treatment on our patients.

Surgery is deemed the only curative technique for pancreatic cancer. Unfortunately, more than 80% of patients who present with the disease cannot be cured by resection.

The literature reports median survival for resectable patients on the order of 19 months, with a 20% 5 year survival rate. For patients unable to undergo surgical resection, the median survival in the literature is approximately 11 months. In the absence of the proposed protocol, this patient population would be treated as per the standard of care for locally advanced non-metastatic surgically unresectable pancreatic malignancies, which would include a combination of chemotherapy and radiation therapy. The anticipated Grade 4 and above toxicity would be approximately 3-5% from this regimen. The rate of G 4 and above toxicity is not known with the use of this neoadjuvant regimen, and, therefore, this constitutes the major risk associated with this protocol therapy. The associated benefit, however, is the anticipated improvement in median survival that these patients may derive from the ability to successfully undergo surgical resection. A secondary proposed benefit is the potential for reduction in the treatment associated toxicity with this altered multimodality schedule when compared to traditional multimodality care or non-surgical care of locally advanced pancreatic malignancy.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed adenocarcinoma of the pancreas
* Resectable or potentially resectable disease based on the following imaging criteria performed < 4 weeks from study entry and as determined by local review (Cooper radiologist)

  * No extrapancreatic extension to nearby organs (ie; small bowel)
  * No SMV/PV >180 degree involvement and/or reconstructable (as determined by Surgeon) occlusion
  * No SMA Abutment TVI<180 degrees
  * No Celiac trunk abutment Total volume involved < 180 degrees
  * Note that both resectable and potentially resectable patients are eligible
* ECOG ≤ 2
* Adequate hematologic and end organ function as defined by

  * Hepatic transaminase levels < 3 x normal
  * Total bilirubin < 5 mg/dl (if stented)
  * Serum creatinine level < 1.6 mg/dl
  * Absolute neutrophil count > 1,500cells/mm3
  * Platelet count > 100,000 cells/mm3
* Medical status suitable for consideration of major pancreatic surgery
* Age >18 years
* Women of childbearing age and male participants must practice adequate contraception (hormonal or barrier method of birth control; abstinence) prior to and throughout study treatment.
* Life expectancy > 3 months
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Prior invasive malignancy within 5 years other than pancreatic adenocarcinoma
* Prior radiotherapy to the upper abdomen
* Severe comorbidity rendering a candidate ineligible for surgical resection
* Local, regional or distant extrapancreatic disease
* Patients of childbearing age who are unwilling or unable to practice contraception
* Failure to meet any of the above eligibility criteria
* Inability to undergo MRI with contrast for treatment planning
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients may not be receiving any other investigational nor commercial agents with therapeutic intent to treat pancreatic cancer while on this trial.
* unresectable pancreatic cancer based on the following imaging criteria performed < 4 weeks from study entry and as determined by local review (Cooper radiologist)

  * Extrapancreatic extension to nearby organs (ie; small bowel)
  * SMV/PV >180 degree involvement and/or reconstructable (as determined by Surgeon) occlusion
  * SMA Abutment TVI<180 degrees
  * Celiac trunk abutment Total volume involved < 180 degrees
  * Distant metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2013-01; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
percentage of subjects who successfully undergo pancreaticoduodenectomy | 2 months
  Evaluate the percentage of subjects who successfully undergo pancreaticoduodenectomy

SECONDARY OUTCOMES:
Overall Survival | 6 months, 1 year, 5 years
Tumor response per RECIST 1.1 | 2-8 months
Quality of Life | 2-8 months
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- MD Anderson Cancer Center at Cooper, Camden, New Jersey, United States